CLINICAL TRIAL: NCT00978081
Title: Photodynamic Therapy for Premalignant and Early Stage Head and Neck Tumors
Brief Title: Photodynamic Therapy in Treating Patients With Premalignant or Early Stage Head and Neck Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000650536; UPCC-18308; IRB #809093; NCT01019954 (obsolete NCT alias)
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Head and Neck Cancer; Precancerous Condition
Keywords: precancerous condition; stage 0 hypopharyngeal cancer; stage 0 laryngeal cancer; stage 0 lip and oral cavity cancer; stage 0 nasopharyngeal cancer; stage 0 oropharyngeal cancer; stage 0 paranasal sinus and nasal cavity cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Precancerous Conditions; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms | interventions — Aminolevulinic Acid

ARMS (2):
- Arm I (Experimental): Patients receive oral aminolevulinic acid and then undergo continuous photodynamic therapy 4-6 hours later.
  Interventions: Drug: aminolevulinic acid hydrochloride
- Arm II (Experimental): Patients receive aminolevulinic acid as in arm I and then undergo fractionated photodynamic therapy 4-6 hours later.
  Interventions: Drug: aminolevulinic acid hydrochloride

INTERVENTIONS:
Drug: aminolevulinic acid hydrochloride — Patients undergo continuous or fractionated photodynamic therapy.

SUMMARY:
RATIONALE: Photodynamic therapy uses a drug that becomes active when it is exposed to a certain kind of light. When the drug is active, tumor cells are killed.

PURPOSE: This randomized phase I trial is studying the side effects and best dose of photodynamic therapy in treating patients with premalignant or early stage head and neck tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the toxicities associated with aminolevulinic acid-mediated photodynamic therapy when administered continuously or in fractionated doses in patients with premalignant or early stage head and neck lesions.

Secondary

* To assess the efficacy of this regimen in these patients.

OUTLINE: This is a dose-escalation study of photodynamic therapy. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral aminolevulinic acid and then undergo continuous photodynamic therapy 4-6 hours later.
* Arm II: Patients receive aminolevulinic acid as in arm I and then undergo fractionated photodynamic therapy 4-6 hours later.

After completion of study therapy, patients are followed up at 1 month, every 3 months for 2 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following within the past 3 months:

  * Erythroplakia with dysplasia
  * Severe dysplasia
  * Carcinoma in situ of the head and neck for which standard therapy is not indicated, according to any of the following:

    * Medical condition that precludes surgery
    * Lesions that cannot be completely resected based on size or location
    * Significant functional morbidity would be anticipated with further surgery
    * Refused standard therapy after the treatment has been discussed and offered
* No invasive squamous cell carcinoma of the head and neck

PATIENT CHARACTERISTICS:

* ECOG performance status of 0-2
* Platelet count ≥ 100,000/mm^3
* Total bilirubin ≤ 2 times upper limit of normal (ULN)
* AST or ALT ≤ 2 times ULN
* Alkaline phosphatase ≤ 2 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior chronic liver disease or cirrhosis of the liver
* No porphyria or hypersensitivity to porphyrins
* No significant cardiovascular history that, in the opinion of a cardiologist, would deem the patient at risk for hypotension that may occur with oral administration of aminolevulinic acid (Levulan®)
* No prior adverse reaction to ondansetron or lorazepam

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | One year
Maximum tolerated dose | 90 days

SECONDARY OUTCOMES:
Response rate | One year
Duration of response | One year
Time to progression | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ahn, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials